#### INDIANA UNIVERSITY INFORMED CONSENT STATEMENT FOR RESEARCH

# Treating Insomnia to Reduce Inflammation in HIV: A Pilot Trial Version 4.0; Protocol#10288

Supported by a grant from the National Institutes of Health (Grant # 1R21MH127206)

## **ABOUT THIS RESEARCH**

You are being asked to participate in a research study. Scientists do research to answer important questions which might help change or improve the way we do things in the future.

This consent form will give you information about the study to help you decide whether you want to participate. Please read this form, and ask any questions you have, before agreeing to be in the study.

#### TAKING PART IN THIS STUDY IS VOLUNTARY

You may choose not to take part in the study or may choose to leave the study at any time. Deciding not to participate, or deciding to leave the study later, will not result in any penalty or loss of benefits to which you are entitled, and will not affect your relationship with your doctors.

## WHY IS THIS STUDY BEING DONE?

The purpose of this study is to determine if treating insomnia, or lack of adequate sleep, in people who are HIV-positive will reduce inflammation in the body. HIV-positive people have greater body inflammation than those without HIV, which leads to a higher chance of developing serious medical conditions in the future, such as heart attacks, kidney failure, dementia, and bone fractures. This greater inflammation in people with HIV is due to many factors, one of which may be insomnia. So by reducing insomnia and helping people with HIV sleep better, there may also be benefits to reducing body inflammation and reduce the chances of having other serious medical problems in the future.

You were selected as a possible participant because you are at least 18 years old, have insomnia, and already are receiving antiretroviral therapy with viral loads (amount of HIV in the bloodstream) that are less than 75 copies per milliliter, or less than 75 HIV virus particles in a milliliter of blood. Women who are pregnant or are breastfeeding are not allowed into this study.

The study is being conducted by Dr. Samir Gupta of the Department of Medicine at the Indiana University School of Medicine and by Dr. Jesse Stewart of the Department of Psychology at the Indiana University-Purdue University-Indianapolis. The study is funded by the National Institutes of Health.

## **HOW MANY PEOPLE WILL TAKE PART?**

If you agree to participate, you will be one of 50 people in Indianapolis to enter the trial.

# WHAT WILL HAPPEN DURING THE STUDY?

This study will compare an interactive, internet-based insomnia treatment program called SHUTi with an education program on better sleep practices. You will be randomly assigned, like a flip of a coin, to one of these two sleep treatment programs. If you agree to be in the study, you will be asked to participate in one Screening Visit, one Entry Visit, another study visit 12 weeks later, and then another study visit 24 weeks after the Entry Visit. If you are chosen to take part in SHUTi, you will be asked to complete an additional six sessions (one per week) over the internet to receive this insomnia

treatment. If you are chosen to receive education on better sleep habits, then our study team will call you to coach you on best ways to improve your sleep.

Because this study involves using a computer, it is important for you to tell us if you have difficulty reading print on a screen. If you cannot use a computer (laptop or desktop) or cannot read and understand instructions on a computer, then you cannot participate in this study.

If you agree to be in the study, you will do the following things at the following study visits:

# Screening Visit

To determine if you qualify for this study, we may first call you on the telephone. With your verbal consent, we will ask if you might wish to participate and if your sleep troubles are severe enough to enter the study. We will use a standard set of questions regarding insomnia to determine if you qualify. We may also ask more about your medical history to make sure you can safely enter the study. If you have had an HIV viral load test done recently, and if it appears you otherwise qualify, we will schedule an Entry Visit appointment with you. If you have not had a recent HIV viral load test, then we will ask you to come into the Infectious Diseases Research Clinic at the Fifth Third Office Building on the Eskenazi Health campus to have this blood test done. The amount of blood to be taken is one teaspoon. If your viral load is lower than 75 copies, then we will schedule the Entry Visit with you.

## **Entry Visit**

The Entry Visit will take no longer than two hours and will take place at the Infectious Diseases Research Clinic at the Fifth Third Office Building on the Eskenazi Health campus. At this visit, we will ask you about your medical and psychiatric history and the medications you take. We will also review your medical records to document your diagnoses and laboratory results as obtained in the clinic. We will measure your height, weight, temperature, blood pressure, and heart rate. You will then be asked to complete a series of surveys related to your sleep, mood, physical activity, fatigue, usual activities, alcohol use, tobacco use, and other substance use. If you are a woman who could become pregnant, we will do a urine pregnancy test. If we find you are pregnant, then your participation in this study will end. We will also do blood tests to check for levels of body inflammation, HIV viral load, and CD4 count (the measure of your immune system affected by HIV). The amount of blood to be taken is no more than 2 tablespoons.

At this time, you will be randomly assigned to either SHUTi or sleep education. Your primary HIV caregiver will be notified about the result of this randomization.

## Entry Visit Follow-Up Call

Between 1 and 14 days after your Entry Visit, a trained research assistant will contact you to complete a sleep disorders interview over the phone. This call is expected to take approximately 20 minutes.

## The Insomnia Treatments Used in This Study

If you are assigned to receive the study insomnia treatment called SHUTi, you will have the opportunity to complete six 40-minute therapy sessions, one per week. These sessions will take place at Dr. Stewart's office on the IUPUI campus, the Infectious Diseases Research Clinic at Eskenazi Hospital, or a location selected by you where you can access a computer with internet, such as your home, your work, a family member's/friend's home, or a public library. Your preference will determine the location

of the SHUTi sessions. The SHUTi sessions will be performed between the Entry Visit and the Week 12 Visit. If you do not have internet access already, we will loan you a tablet computer with free internet connection for use during this study. You must return this computer at the Week 12 Visit.

The insomnia treatment is an interactive computer program; therefore, you will not be meeting face-to-face with a therapist. Through completing the sessions on a computer, you will learn techniques that have been shown to improve insomnia in other types of patients. These techniques include learning what causes your lack of sleep, how to improve your chances of better sleep, and how to avoid those things that cause your poor sleep. Please note that this program may be more effective in treating your insomnia if you are able to complete more of these sessions. You will then be given homework to complete before the next session; homework is to help you achieve better sleep.

As part of the SHUTi program, you will be asked to enter information regarding your particular sleep problem. This will help SHUTi make an individual treatment plan for you. You will not enter any information that can identify you other than the email address you choose to use to receive messages (such as reminders) from the program. You will only be known to the program by a unique identification number.

If you are assigned to the sleep education group of the study, our study team will provide you access to an internet-based sleep education program that will inform you about ways to improve your sleep. You will not enter any information that can identify you other than the email address you choose to use to receive messages (such as reminders) from the program. We will also email or mail you a list of places you can get more information and help about improving your sleep. Our study team will also call you once per month to see if your insomnia symptoms are improving; if not, then we will notify your HIV provider who may provide additional counselling or treatment for poor sleep.

Regardless of which treatment group you are assigned, you will also complete sleep diaries electronically for the 14 days prior to the Week 12 and Week 24 study visits.

## Week 12 Visit

You will then be asked to return to the Infectious Diseases Research Clinic in approximately 12 weeks after the Entry Visit. This visit will take no more than 2 hours. We will review your medical records and medications again, especially if your doctor has started any new insomnia treatments since your last visit. Your blood pressure, heartrate, temperature, and weight will also be measured again. We will also ask you to complete the same surveys regarding your sleep, mood, physical activity, fatigue, usual activities, alcohol use, tobacco use, and substance use. If you are a woman who could become pregnant, we will do a urine pregnancy test. If we find you are pregnant, then your participation in this study will end. We will also do blood tests to check for levels of body inflammation, HIV viral load, and CD4 count (the measure of your immune system affected by HIV). The amount of blood to be taken is no more than 2 tablespoons.

## Week 24 Visit

You will then be asked to return to the Infectious Diseases Research Clinic in approximately 24 weeks after the Entry Visit (or about 12 weeks after the Week 12 Visit). This visit will take no more than 2 hours. We will review your medical records and medications again, especially if your doctor has started any new insomnia treatments since your last visit. Your blood pressure, heartrate, temperature, and

weight will also be measured again. We will also ask you to complete the same surveys regarding your sleep, mood, physical activity, fatigue, usual activities, alcohol use, tobacco use, and substance use. If you are a woman who could become pregnant, we will do a urine pregnancy test. If we find you are pregnant, then your participation in this study will end. We will also do blood tests to check for levels of body inflammation, HIV viral load, and CD4 count (the measure of your immune system affected by HIV). The amount of blood to be taken is no more than 2 tablespoons. So overall, the amount of blood that will be taken will be no more than 6 tablespoons.

At this time your participation in the study will be completed.

## WHAT ARE THE RISKS OF TAKING PART IN THE STUDY?

While participating in the study, the risks, side effects, and/or discomforts include:

# Risks of possibly experiencing emotional discomfort when completing surveys

The surveys will be given in private settings. You may choose not to answer any questions that make you feel uncomfortable.

# The risks of possible loss of confidentiality

We will not tell anyone other than your main HIV caregiver that you are taking part in this study. All of your information will be identified with a coded number and without any personal identifying information. All test results will be locked in a cabinet and restricted.

If you choose to undergo the SHUTi insomnia treatment sessions at Dr. Stewart's office or the Infectious Diseases Research Clinic, you will be in a private location where others, besides the study team members, cannot see you. But please note that if you choose to undergo the SHUTi treatment sessions in a public location, others around you may see that you are viewing an online insomnia treatment program. We will give you ear bud headphones, if you do not already have headphones, if you choose to complete the treatment sessions at a public location.

## The risks of drawing blood

There are small risks in blood draws as part of this study, which include pain, bruising, infection, and damage to the veins in your arm.

## Suicidal thoughts

Because this study may involve people who have depression, some participants may report thoughts of being better off dead or of hurting themselves. This could happen during a phone call or an in-person visit. IF this occurs, our protection plan will be used. You will first be asked a series of questions. If it is determined that immediate care is needed, the study team will contact Dr. Stewart and/or Dr. Gupta to determine the right course of action. If we believe that you are in imminent danger of harm, we will have to report it, potentially to authorities, including the police, for your own protection. We may contact your primary doctor, your primary HIV caregiver, and your HIV social worker or care coordinator. We may also consult with the LifeCare clinic psychiatrist or with Midtown Community Mental Health Center and escort you to the Crisis Intervention Unit at Eskenazi Health Hospital.

If you prematurely terminate a phone call after reporting suicidal thoughts, the study doctors will be notified to determine the right course of action. We will try to contact you back to obtain additional

information. If it is determined that immediate care is needed and that you are in imminent danger of harm, we will have to report it, potentially to authorities, including the police, for your own protection. We may contact your primary doctor, your primary HIV caregiver, and your HIV social worker or care coordinator. We may also consult with the LifeCare clinic psychiatrist or with Midtown Community Mental Health Center and refer you to the Crisis Intervention Unit at Eskenazi Health Hospital.

We may also then decide in this situation that it is important for your own safety to end your participation in this trial.

# Are there risks if I get pregnant during the study?

No. But if you do become pregnant, then we will remove you from further study participation as pregnancy affects the way we measure inflammation in this trial.

## WHAT ARE THE POTENTIAL BENEFITS OF TAKING PART IN THE STUDY?

You may receive no direct benefit from participating in this study. However, you may receive benefits if the insomnia treatment program improves your sleep and reduces the amount of body inflammation. Information learned from this study may help others who have HIV.

#### ALTERNATIVES TO TAKING PART IN THE STUDY:

Instead of being in the study, you have the option not to participate and choose to seek other types of insomnia treatment through your HIV caregiver. The most common alternative treatments for insomnia are medications and psychotherapy. If you choose not to participate, your decision will not affect your regular medical care or your relationship with the study doctor.

## WILL I RECEIVE MY RESULTS?

We may learn things about you from the study activities which could be important to your health or to your treatment. If this happens, this information will be provided to you. We might learn about your HIV status or if you have depressed mood. We will provide you these results if they are abnormal or worrisome. If you wish to see these results even if normal, we will provide you a copy. You may need to meet with professionals with expertise to help you learn more about your results. However, the study team/study will not cover the costs of any follow-up consultations or actions.

# **HOW WILL MY INFORMATION BE PROTECTED?**

Efforts will be made to keep your personal information confidential. We cannot guarantee absolute confidentiality. Your personal information may be disclosed if required by law and/or to individuals or organizations that oversee the conduct of research studies. No information which could identify you will be shared in publications about this study.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use any information, documents, or specimens that could identify you in any legal action or lawsuit unless you say it is okay.

However, there are some types of sharing the Certificate does not apply to. The Certificate does not stop reporting required by federal, state, or local laws, such as reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate does not stop a government agency who is funding research from checking records or evaluating programs. The

Certificate also does not prevent your information from being used for other research when allowed by federal regulations. The Certificate also does not stop sharing of information required by the Food and Drug Administration (FDA).

Researchers may release information about you when you say it is okay. For example, you may still give them permission to release information to insurers, medical providers, or others not connected with the research.

A description of this clinical trial is available on <u>ClinicalTrials.gov</u> (Record # NCT04721067) as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

## WILL MY INFORMATION BE USED FOR RESEARCH IN THE FUTURE?

Information or specimens collected from you for this study may be used for future research studies or shared with other researchers for future research. If this happens, information which could identify you will be removed before any information or specimens are shared. Since identifying information will be removed, we will not ask for your additional consent.

We may use your blood specimens to learn more about how insomnia affects HIV and body inflammation. We will store all blood specimens using only your study code and keep them in the research freezers of Dr. Gupta. The research freezer is kept in a locked room in the R3 Research Building at Indiana University School of Medicine. Only Dr. Gupta and his study team have access to the research freezers in which your blood specimens will be stored. To protect you against the risks of loss of confidentiality, all samples will be marked with a unique code number. This information will be stored in an anonymous fashion in two different secured computer databases; one containing the sample codes and the other with your information (such as age, sex, ethnic group, health conditions, etc.) to maximize confidentiality.

# **Making Your Choice**

Blood and urine samples will be collected as part of your screening and/or during the study period. We will not obtain DNA or other kinds of genetic samples. Please read each sentence below and think about your choice. After reading each sentence, circle or check "Yes" or "No" and add your initials next to the choice. No matter what you decide it will not affect your care or your ability to participate in this study. If you have any questions, please talk to your doctor or nurse or call our Institutional Review Board, whose contact information can be found on the next page.

You retain (keep) the right to have any remaining sample material destroyed at any time by contacting the investigator. The investigator is responsible for the destruction of the sample at your request. However, any previously collected data from your sample cannot be destroyed.

| | learn more about how to treat health problems. | |
|---|---|---|
| | YES | NO |
| 2. | Someone can contact me in the future to ask me to take part in more research. | |
| | YES | NO |

1. My sample(s) may be kept for a period of up to 20 years or more for use in future research to

## WILL I BE PAID FOR PARTICIPATION?

You will be compensated \$50 after completing the Entry Visit, \$50 after completing the Week 12 Visit, and \$75 after completing the Week 24 Visit. There is no compensation for the Screening Visit. Payment will be in the form of a pre-paid gift card or by a refillable gift card.

For any in-person visit (Screening, Entry, and Week 12 and Week 24), you may be eligible for no-cost transportation from your home to and from the clinic via Uber Health. Please discuss this with the study staff to make travel arrangements.

## WILL IT COST ME ANYTHING TO PARTICIPATE?

There is no cost to you for taking part in this study.

## WHO WILL PAY FOR MY TREATMENT IF I AM INJURED?

In the event of physical injury resulting from your participation in this study, necessary medical treatment will be provided to you and billed as part of your medical expenses. Costs not covered by your health care insurer will be your responsibility. Also, it is your responsibility to determine the extent of your health care coverage. There is no program in place for other monetary compensation for such injuries. However, you are not giving up any legal rights or benefits to which you are otherwise entitled.

## WHAT FINANCIAL INTEREST DOES THE RESEARCHER HAVE?

Neither Dr. Gupta nor Dr. Stewart have any financial interests in the outcomes of this study.

## WHO SHOULD I CALL WITH QUESTIONS OR PROBLEMS?

For questions about the study or a research-related injury, you may call the Infectious Diseases Research Clinic at 317-278-2945. You may also contact the researchers, Dr. Samir Gupta at 317-274-7926 or Dr. Jesse Stewart at 317-274-6761. After business hours (8:00 AM-4:00 PM from Monday-Friday), please call the on-call Infectious Diseases physician <u>for Indiana University Hospital</u> at 317-944-5000.

For questions about your rights as a research participant, to discuss problems, complaints, or concerns about a research study, or to obtain information or to offer input, please contact the IU Human Subjects Office at 800-696-2949 or at irb@iu.edu.

## **CAN I WITHDRAW FROM THE STUDY?**

If you decide to participate in this study, you can change your mind and decide to leave the study at any time in the future. No risks are involved by leaving the study. If you decide to withdraw, please contact the study coordinator or Dr. Samir Gupta. Your future medical care will not be affected by your decision to leave the study.

The study researchers may need to take you off the study without your permission if they feel it is not in your best interest for you to participate.

#### **PARTICIPANT'S CONSENT**

In consideration of all of the above, I give my consent to participate in this research study. I will be given a copy of this informed consent document to keep for my records. I agree to take part in this study.

| Participant's Printed Name: | |
|-------------------------------------------|-------|
| Participant's Signature: | Date: |
| Printed Name of Person Obtaining Consent: | |
| Signature of Person Obtaining Consent: | Date: |